CLINICAL TRIAL: NCT01080677
Title: Randomized Double-Blind Study to Evaluate the Dose-Related Efficacy and Safety of Caffeine/Propranolol in the Treatment of Acute Migraine
Brief Title: Caffeine/Propranolol Intervention for Acute Migraine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, S. Charles Cho, Principle Investigator, Stanford University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: SU-02112010-4963; 7011 (Other Grant/Funding Number: Palo Alto Institute/Stanford University)
Record Dates: First submitted 2010-03-02; First posted 2010-03-04 (Estimated); Results first posted 2017-02-24 (Actual); Last update posted 2017-02-24 (Actual); Status verified 2017-01

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Participants will receive placebo to match caffeine/propranolol (single dose)
  Interventions: Drug: placebo
- Low dose (Experimental): Participants will receive caffeine/propranolol 400/40 mg combination tablet (single dose)
  Interventions: Drug: caffeine/propranolol combination tablet
- High dose (Experimental): Participants will receive caffeine/propranolol 1000/40 mg combination tablet (single dose)
  Interventions: Drug: caffeine/propranolol combination tablet

INTERVENTIONS:
Drug: caffeine/propranolol combination tablet — caffeine/propranolol combination tablet administered orally once daily
  Arms: High dose; Low dose
Drug: placebo — placebo to match caffeine/propranolol combination tablet administered orally once daily
  Arms: Placebo

SUMMARY:
This is a research study to assess the safety of caffeine/propranolol at different dose levels. We want to find out what effects, good and/or bad, it has on patients and their migraines.

DETAILED DESCRIPTION:
There will be a screening exam to find out if potential subjects are eligible to be in the main part of the study. Screening will include obtaining demographics, migraine history, migraine characteristics, verification that subjects's migraine satisfies the International Headache Society criteria, migraine medication history with success and failure rates, and medical history.

If a subject is female, we will need to confirm to the extent medically possible that they are not pregnant. Female subjects must agree to have a urine pregnancy test done before beginning this research study. If a subject is a woman who is able to become pregnant, it is expected that they will use an effective method of birth control to prevent exposing a fetus to a potentially dangerous agent with unknown risk. They must accept the risk that pregnancy could still result despite the responsible use of reliable method of birth control.

They agree to notify Dr. Cho as soon as possible of any failure of proper use of your birth control method, or if you become pregnant, either of which may result in your being withdrawn from the study.

Subjects will also undergo a liver function test as well as an EKG to make sure they are eligible for the study.

Once subject eligibility has been determined, they will be randomized to one of 3 study groups described below. Neither the subjects nor the doctor can choose which group subjects will be in nor will subjects or their doctor know which group subjects are in. They will have a one in three chance of being placed in any group. Two groups will be active treatment with either 400 mg caffeine and 40 mg propranolol or 1000 mg caffeine and 40 mg propranolol. The third group will be a placebo group with no active medication.

Subjects will then be given a study kit, which includes caffeine/propranolol or placebo oral medication, a treatment booklet, migraine headache diary, pen and stopwatch. The study coordinator will then instruct them in the accurate method of diary completion and use of the oral medication or placebo pill. Their final visit will be scheduled within 60 days of enrollment.

They will be instructed to treat one moderate or severe migraine attack with the study medication. They will be instructed to take study medication at aura onset in the presence of another adult.

In the absence of any aura, they will be instructed to take study medication at headache onset. Another adult should be present when taking the study medication to ensure safety. In the event that the migraine occurs while they are alone, the subjects are instructed not to take the study medication and to wait for the next headache when adult supervision is available. They will not be allowed to use any non-steroidal,anti-inflammatory drugs such as ibuprofen or naproxen sodium, non-prescription analgesics such as acetaminophen or aspirin, narcotic analgesics such as oxycontin, oxycodone, triptan or ergotamine medication or derivatives (Cafergot®, D.H.E., 45®[dihydroergotamine mesylate], Efcaf®, Ergomar®, Ergostat®, Migranal®, Nasal Spray, Sansert®[methysergide], or Wigraine®) within 24 hours prior to dosing with the study medication. Subjects will also be instructed not to use any caffeine such as coffee, tea, caffeine containing sodas, or caffeine containing medications (Cafcit®, Caffedrine®, Enerjets, Lucidex, No Doz® Maximum Strength, Vivarin®) within 6 hours prior to dosing with the study medication.

Subjects will record the severity of their headache and associated symptoms at baseline and 15, 30, 45, 60, and 120 minutes after dosing. If the migraine does not resolve or worsens after 2 hours, they will be allowed to take #rescue medication# as prescribed by their physician. Subjects will continue to record the severity of their headache and associated symptoms for 4, 12, and 24 hours after initial dosing. Following the last entry in the subject diary at 24 hours, they will be asked to complete a treatment satisfaction questionnaire. They will also be asked to contact Dr. Cho#s office to review their diary completion and to confirm the date of their final visit.

If subjects have not called to report a migraine within a month (±7 days) of enrollment, Dr. Cho or someone from his research staff will call them to determine if they have treated a migraine. If a migraine was treated, Dr. Cho or the study staff will interview them to determine if the diary has been appropriately completed and to ensure that adequate information has been recorded. Their final visit will be confirmed and should occur within 30 days of the treated migraine. If they have not treated a migraine with the study medication within the first 30 days of enrollment, their final visit will be rescheduled within 60 days of your enrollment date (± 7 days).

At the final visit, the study coordinator will review their subject diary for completeness and accuracy. All study materials will need to be returned at this visit. Subjects will then have a second EKG to make sure the medication didn't have any negative effects on their cardiac function. Subjects will be given a voucher to pay for parking expenses. In addition, there will be a data safety monitoring unblinding event after the first 15 patients have completed the study. All serious and non-serious adverse events will be analyzed regardless of the investigators' assessments of causality. Adverse events that result in death, hospitalization, permanent disability or threat to life are classified as serious. The Medical Dictionary of Regulatory Activities (MedDRA) will be used to categorize reported adverse events. Someone who is not directly related to the research team will conduct the safety monitoring.

If there are any serious adverse events during the study, the study will be discontinued.

ELIGIBILITY:
Inclusion Criteria:1. Subject has a minimum 12-month migraine history that the investigator determines meets the International Headache Society (IHS) Migraine Diagnostic Criteria for migraine with or without aura 2. Subject is between 18-50 years of age. 3. Subject experiences an average of 2-8 migraines per month. 4. If on preventive migraine therapy, medication regimen has been stable for 30 days and will remain stable for the duration of participation.

5. Subject is able to communicate adequately and comply with the requirements of the study as determined by the investigator.

6. Subject is able to read and understand the informed consent written in English and voluntarily consents to sign the informed consent form.

Exclusion Criteria:1. Subject#s age of migraine onset is greater than 50 years. 2. Subject has more than 6 non-migraine headache days per month. 3. Subject has less than 48 hours of freedom from headache between attacks of migraine.

4. Subject meets the criteria for complicated and/or brainstem migraines. 5. Subject is pregnant or lactating. 6. Subject has history of alcohol or drug abuse within the past 2 years. 7. Subject has existing systolic blood pressure < 100mm Hg, existing systolic blood pressure > 150mm Hg, and or heart rate <50 beats per minute.

8. Subject has heart block greater than 1st degree without a functioning pacemaker 9. Subject has a history of tachyarrythmias 10. Subject has uncompensated congestive heart failure (CHF) 11. Subject has severe chronic obstructive pulmonary disease or severe asthma. 12. Subject has consumed caffeine within 6 hours. 13. Subjects with existing generalized anxiety disorder (GAD) and/or panic disorder.

14. Subjects with existing severe hepatic and/or renal insufficiency. 15. Subjects with existing Raynaud#s disease. 16. Subject is participating in another clinical trial during or within 30 days prior to study enrollment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2007-01; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: S. Charles Cho, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo to match caffeine/propranolol (single dose)
- Low Dose: Participants received caffeine/propranolol 400/40 mg combination tablet (single dose)
- High Dose: Participants received caffeine/propranolol 1000/40 mg combination tablet (single dose)
Period: Overall Study
Arm/Group | Placebo | Low Dose | High Dose
Started | 20 | 20 | 20
Completed | 20 | 20 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Thirty females, thirty males, agews ranged from 18-50 years old. All had an established history of migraines for at least 1 year. All met the diagnostic criteria of the International Classification of Headache Disorders.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Low Dose | High Dose | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 15 | 45
  >=65 years | 5 | 5 | 5 | 15
Gender [Count of Participants; unit: Participants]
  Female | 10 | 10 | 10 | 30
  Male | 10 | 10 | 10 | 30
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 20 | 60

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting Pain Relief at 2 Hrs Post First Administration of Caffeine/Propranolol (Defined as a Decrease in Headache Pain Intensity From Severe or Moderate Headache Pain at Baseline to Mild or no Pain at 2 Hrs)
Time Frame: 2 hours
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Low Dose | High Dose
Number analyzed (Participants) | 20 | 20 | 20
percentage of participants | 10 | 45 | 60

2. Secondary Outcome: Percentage of Participants Pain Free at 2 Hrs Post First Administration of Caffeine/Propranolol
Time Frame: 2 hours
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Low Dose | High Dose
Number analyzed (Participants) | 20 | 20 | 20
percentage of participants | 0 | 20 | 35

3. Secondary Outcome: Percentage of Participants Experiencing at Least One Adverse Event of Interest
Description: Adverse events may have included abdominal pain, flushing, dizziness, insomnia, or anxiety
Time Frame: 24 hours
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Low Dose | High Dose
Number analyzed (Participants) | 20 | 20 | 20
percentage of participants | 10 | 25 | 50

4. Secondary Outcome: Percentage of Participants With Treatment Satisfaction
Description: Following up to 24 hours after treatment, participants were asked to report whether they were satisfied with level of pain relief provided by treatment
Time Frame: 24 hours
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Low Dose | High Dose
Number analyzed (Participants) | 20 | 20 | 20
percentage of participants | 5 | 40 | 80

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Placebo | Low Dose | High Dose
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 4/20 | 5/20 | 5/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=20) | Low Dose (N=20) | High Dose (N=20)
abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
insomnia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
flushing (General disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No